CLINICAL TRIAL: NCT03569956
Title: The Impact of the 556 Razor Technology and of a Regimen of the 556 Razor Technology With Pre-Shave Gel and Brush on Shaving Satisfaction in Males With Skin Irritation From Shaving
Brief Title: Shaving Satisfaction in Males With Skin Irritation From Shaving
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00051291
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pseudofolliculitis Barbae
Keywords: Razor bumps; Skin Irritation; Shaving
MeSH Terms: conditions — pseudofolliculitis barbae

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into two groups: the Razor group of 20 subjects, and the Regimen group of 20 subjects. In the Razor group, subjects will use the 556 Razor with their regular shaving products, and shave at least 5 or more times per week. In the Regimen group, subjects will use the 556 Razor, Pre-Shave Gel, Cleansing brush and Shaving Gel, and shave at least 5 or more times per week. All subjects will be given the 556 Razors during the 12-week study. The Regimen group will also be given the Pre-Shave Gel, Cleansing Brush, and Shaving Gel.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Razor Group (Active Comparator): Subject will use the 556 razor with regular shaving products, and shave at least 5 or more times per week
  Interventions: Other: 556 Razor
- Regimen (Experimental): Subject will use the 556 razor with the Pre-shave Gel, Cleaning Brush, and Shaving Gel and shave at least 5 or more times per week.
  Interventions: Other: 556 Razor

INTERVENTIONS:
Other: 556 Razor — In the Razor group, subjects will use the 556 Razor with their regular shaving products, and shave at least 5 or more times per week. In the Regimen group, subjects will use the 556 Razor, Pre-Shave Gel, Cleansing brush and Shaving Gel, and shave at least 5 or more times per week. All subjects will be given the 556 Razors during the 12-week study. The Regimen group will also be given the Pre-Shave Gel, Cleansing Brush, and Shaving Gel.

SUMMARY:
The purpose of this research study is to evaluate the improvement in overall shave satisfaction, the appearance of skin irritation from shaving, and the razor related inflammation of the hair follicles when using a new razor technology in a regular shaving regimen as well as a new razor technology in a shaving regimen that includes a pre-shave gel, cleansing brush and shaving gel.

DETAILED DESCRIPTION:
A secondary objective is to show improvement in the satisfaction of the shaving experience, symptoms such as bumps and irritation, and quality of life (QOL), when adding the 556 Razor, or the 556 Razor with a regimen of pre-shave gel, cleansing brush, and shave gel to the shaving regimen of males with shaving skin irritation. Shaving irritation severity will be correlated to shave satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Males with at least a two year history of the symptoms of skin irritation from shaving.
2. Must be age 20-60 years of age (inclusive).
3. Must wet shave using just a prep and blade razor at least 3 or more times per week, and be willing to shave at least 5 times per week during the study
4. Must have Mild to moderate symptoms of skin irritation from shaving based on IGA rating scales. There must be the presence of some razor bumps but there are no lesion count inclusion requirements.

Exclusion Criteria:

1. Changes in the use of systemic (oral antibiotics) within the last 4 weeks. Stable use of oral antibiotics for any condition are allowed
2. Changes in the use of topical prescriptions
3. Individuals who do not wet shave with a bladed razor, or who use electric shavers.
4. Individuals who have removed a beard within last two months.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Shaving Satisfaction and Appearance score | Baseline, Week 4, Week 8, Week 12
  Shaving Satisfaction and Appearance will be captured by the subject during 12 week time frame to document changes in severity and appearance and assessed by the Patient Global Severity Assessment. The score range is 0-30. The lower the scores; the better the outcome.
Change in Investigator Global Severity Assessment (IGA) score | Baseline, Week 4, Week 8, Week 12
  Disease severity will be assessed Investigator Global Severity Assessment (IGA). Appearance will be captured by the PI by using a scale 0 (clear) to 5 (very severe) during the 12 week time frame to document changes in severity and appearance. The score range is 0-5. The lower the scores, the better the outcome.

SECONDARY OUTCOMES:
Disease severity assessed by lesion counts | Baseline, Week 4, Week 8, Week 12
  Disease severity will be assessed by lesion counts of any follicular papules in the beard area (not including acne) pustules, excoriations, hyperpigmentation, and ingrown hairs. Higher scores are indicative of worse outcome because more lesions mean more involvement of the razor bumps and associated inflammation.

OTHER OUTCOMES:
Patient's Global Severity Assessment (PGSA)- satisfaction of shaving experience | Baseline, Week 4, Week 8, Week 12
  Change in the satisfaction of Shaving experience by subjects completing the patients's global severity assessment during the 12 week study. The score range is 0-30. The lower the scores, the better the outcome.
Change in Patient's Global Severity Assessments- skin irritation | Baseline, Week 4, Week 8, Week 12
  Change in skin irritation will be evaluated by subjects by completing the patients's global severity assessment during the 12 week study. The score range is 0-30. The lower the scores, the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J McMichael, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No